CLINICAL TRIAL: NCT02294994
Title: Randomized Controlled Clinical Study to Compare the Efficacy and Safety of Different Dose of Tirofiban in Interventional Treatment of Complex Coronary Artery Disease
Brief Title: Efficacy and Safety of Different Dose of Tirofiban in Interventional Treatment of Complex Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SecondJilinU-1
Record Dates: First submitted 2014-11-16; First posted 2014-11-19 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tirofiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- half dose tirofiban (Experimental): Tirofiban was administered once the wire had crossed the lesion during PCI with a bolus dose of 25 µg/kg of bodyweight, followed by an infusion of 0.075 µg per kilogram per minute for 24 to 36 hours.UFH heparin was administered as a bolus of 100 U/kg before PCI.
  Interventions: Drug: tirofiban
- recommended-dose Tirofiban (Active Comparator): Tirofiban was administered once the wire had crossed the lesion during PCI with a bolus dose of 25 µg/kg of bodyweight, followed by an infusion of 0.15 µg per kilogram per minute for 18 to 24 hours. UFH heparin was administered as a bolus of 100 U/kg before PCI.
  Interventions: Drug: tirofiban
- none tirofiban (Placebo Comparator): Tirofiban was not administered ,UFH heparin was administered as a bolus of 100 U/kg before PCI.
  Interventions: Drug: tirofiban

INTERVENTIONS:
Drug: tirofiban
  Other Names: GPIIb/IIIa inhibitor; aggrastat

SUMMARY:
The aim of the study is to investigate the efficacy and safety different dose of GPIIb/IIIa inhibitor (tirofiban) in interventional treatment of complex coronary artery disease ,which include bifurcation lesion, left main lesion, multiple vessel disease, intracoronary thrombus, SYNTAX score>26,chronic total occlusion disease. The primary endpoint is all-cause mortality. Secondary endpoints are incidence of major bleeding and the rate of site access complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients were recruited from those undergoing PCI with a planned placement of an intracoronary stent
* Including patients with unstable angina pectoris, acute coronary syndrome or NSTEMI
* Experienced ischaemic pain at rest
* Lasting 10 minutes and occurring within 7 days before enrollment
* As well as one of the following: ECG changes: New or presumably new ST-segment depression greater than or equal to 0.1 mV (1 mm), or transient (< 30 minutes) ST-segment elevation greater than or equal to 0.1 mV (1 mm) in at least 2 contiguous leads -Abnormal cardiac enzymes within the 24 hours before enrollment, defined as elevated Troponin I defined as elevated Troponin I (above the normal reference -
* High-risk angiographic features :lesion/anatomy related bifurcation lesion, left main lesion, multiple vessel disease, intracoronary thrombus, SYNTAX score > 26 and chronic total occlusion disease.

Exclusion Criteria:

* Increased bleeding risk: ischaemic stroke within the last year or any previous haemorrhagic stroke, tumour or intracranial aneurysm;
* Recent (<1 month) trauma or major surgery (including bypass surgery);
* Active bleeding
* Unexplained clinically significant bleeding, thrombocytopenia (platelet count < 100 x 109/L) or history of thrombocytopenia with GP IIb/IIIa, heparin or enoxaparin therapy
* Angina from secondary causes such as severe uncontrolled hypertension (systolic blood pressure > 180 mm Hg despite treatment)
* Valvular disease, congenital heart disease, hypertrophic cardiomyopathy, - Thrombolytic therapy within preceding 24 hours
* Receiving antiIIb/IIIa therapy
* Creatinine clearance of <30 mL/min

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical Events | 30 days
  A composite of all cause death, reinfarction, urgent target vessel revascularization, stroke and any bleedings

SECONDARY OUTCOMES:
Net adverse clinical events | 1 year
  a composite of all cause death, any myocardial infarction, any target vessel revascularization, stroke or any bleedings
any bleedings (BARC class) | 30 days
  including all BARC class (class 1-5)
Major adverse cardiac and cerebral events (MACCE) | 30 days and 1 year
  a composite of all cause death, reinfarction, target vessel revascularization or stroke
stent thrombosis | 30 days and 1 year
  by ARC definition

CONTACTS AND LOCATIONS:
Overall Officials: Liu Bin, M.D., Principal Investigator — Jilin University
Locations (1):
- The sencond hospital of Jilin University, Changchun, Jilin, China